CLINICAL TRIAL: NCT05471518
Title: Sex Hormone and Vascular Function in Women With CKD
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3018
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-menopausal women with CKD: Age 18-44 years CKD stage 3-4 (eGFR 15-59 ml/min/1.73m2)
  Interventions: Other: No intervention
- Post-menopausal women with CKD: Age 55-75 years CKD stage 3-4 (eGFR 15-59 ml/min/1.73m2)
  Interventions: Other: No intervention
- Pre-menopausal healthy women: Age 18-44 years Regular menstrual cycle (25-35 d)
  Interventions: Other: No intervention
- Post-menopausal healthy women: Age 55-75 years
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The risk of cardiovascular disease (CVD) is significantly elevated in patients with chronic kidney disease (CKD). Notably, women with CKD commonly experience menstrual disturbances induced by CKD, which may contribute to impaired vascular function and elevated CVD risk. However, most of the literature in the field of nephrology focuses on male patients, and studies on women's vascular health are limited. Moreover, endogenous sex hormones, particularly estradiol, are well-documented to be cardioprotective in women without CKD; however, the role of sex hormones on vascular function in women with CKD remains unclear. The goals of the proposed project are: 1) to evaluate vasuclar function in pre- and post-menopausal women with CKD vs. age-matched healthy women; 2) to evaluate sex hormone concentrations and determine whether they associate with vascular function in the proposed cohort; and 3) to gain mechanistic insight on the association between sex hormones and vascular dysfunction in the proposed cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Pre- (18-44 y) and post-menopausal (55-75 y) women
2. Individuals with CKD including stage 3-4 (eGFR 15-59 ml/min/1.73m2) determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation AND/OR urinary albumin-creatinine ratio (UACR) ≥ 30.
3. Controls must be healthy (free from hypertension, kidney disease, cardiovascular disease, diabetes, and other chronic disease as assessed by self-report, medical history, and screening labs). Premenopausal healthy women must have a regular menstrual cycle (25-35 d).

Exclusion Criteria:

1. Perimenopausal (45-54 y) women
2. Pregnancy, lactation, or less than one year post-partum
3. Use of hormonal birth control methods, hormone replacement therapy, or a levonorgestrel intrauterine device (IUD) insertion for a duration less than 6 months
4. Advanced CKD requiring dialysis
5. History of kidney transplant
6. Use of immunosuppressant medications (unless taking a stable dosage for a quiescent disease in CKD group)
7. Antioxidant and/or omega-3 fatty acid use within the 2 weeks prior to testing
8. Current tobacco or nicotine use or history of use in the last 12 months
9. Marijuana use within 2 weeks prior to testing
10. Uncontrolled hypertension in CKD group (BP >140/90 mmHg)
11. Atrial fibrillation
12. Active infection or antibiotic therapy
13. Hospitalization in the last month

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pre- and post-menopausal women with CKD vs. age-matched healthy women
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation | Baseline
  Flow-mediated dilation of the brachial artery will be performed using ultrasonography and analyzed with a commercially available software package as percent change in diameter from baseline following reactive hyperemia.

SECONDARY OUTCOMES:
Carotid Femoral Pulse Wave Velocity | Baseline
  A transcutaneous custom tonometer [Noninvasive Hemodynamics Workstation (NIHem), Cardiovascular Engineering Inc.] will be used to non-invasively assess carotid femoral pulse wave velocity.
Serum Sex Hormones | Baseline
  Serum sex hormones [follicle-stimulating hormone (FSH), luteinizing hormone (LH), estradiol, progesterone, prolactin, sex hormone binding globulin (SHBG), and anti-mullerian hormone (AMH)] will be measured using chemiluminescent assays.
Urinary Sex Hormones | Baseline
  Urinary sex hormones [follicle-stimulating hormone (FSH), luteinizing hormone (LH), estrone-3-glucuronide (E1c), and pregnanediol-3-glucuronide (Pdg)] will be measured by by chemiluminescent assays using ACS-180 Autoanalyzer.

OTHER OUTCOMES:
Circulating/Urinary Markers of Antioxidant Status/Oxidative stress | Baseline
  Serum TAS, plasma/urinary 8-isoprostane, 8-OHdG will be measured using ELISA.
Circulating Markers of Inflammation | Baseline
  Plasma CRP, IL-1β, IL-6, and TNF-α will be measured using ELISA
Cytokine secretion from lipopolysaccharide(LPS)-stimulated peripheral blood mononuclear cells (PBMCs) | Baseline
  PBMCs will be isolated from heparinized whole blood using Cell Preparation Tube, PBMCs will be cultured with LPS, and supernatants will be harvested after 4-hour stimulation at 37°C. IL-1β, IL-6, and TNF-α in the supernatants will be measured using ELISA.
Distribution of Monocyte Subsets | Baseline
  PBMCs will be stained with fluorescence-labeled antibodies for monocyte (CD14 and CD16) and analyzed using an LSR II flow cytometer.
Ex Vivo Nitric Oxide Production from Human Umbilical Vein Endothelial Cells (HUVECs) | Baseline
  HUVECs will be incubated with basal media supplemented with 10% human serum collected from participants and stained with the fluorescent probe DAF-FM diacetate to detect nitric oxide production production in response to acetylcholine.
Ex Vivo Reactive Oxygen Species Production from Human Umbilical Vein Endothelial Cells (HUVECs) | Baseline
  HUVECs will be incubated with basal media supplemented with 10% human serum collected from participants and stained with the fluorescent probe DAF-FM diacetate to detect reactive oxygen species production in response to acetylcholine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in CKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).